CLINICAL TRIAL: NCT07311304
Title: A Randomized Controlled Trial on the Efficacy of Early Task-Oriented Rehabilitation in Acute Stroke Recovery Compared to Traditional Rehabilitation
Brief Title: Efficacy of Early Task-Oriented Rehabilitation in Acute Stroke Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Asaad Fahmy, Researcher, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Task-Oriented Rehabilitation
Record Dates: First submitted 2025-09-27; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Ischemic Stroke; Hemorrhagic Stroke
Keywords: Task-Oriented Rehabilitation; Early Rehabilitation; Stroke Recovery; Neurorehabilitation; Physical Therapy; Motor Function; Ischemic Stroke; Hemorrhagic Stroke; Randomized Controlled Trial
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Task-Oriented Rehabilitation (Experimental): Participants receive a structured task-oriented rehabilitation program emphasizing functional, goal-directed activities. Examples include upper-limb tasks (reaching, grasping, buttoning, simulated self-care), lower-limb tasks (sit-to-stand, gait training, stair climbing), and balance tasks (carrying a tray, obstacle negotiation). Sessions occur 3-4 times per week, 45-60 minutes each, during hospitalization and continued as outpatient follow-up. Progression is graded by difficulty, repetitions, and patient tolerance.
  Interventions: Behavioral: Task-Oriented Rehabilitation
- Active Comparator: Traditional Physiotherapy Rehabilitation (Active Comparator): Participants receive conventional physiotherapy including stretching, range-of-motion exercises, muscle activation techniques, balance training, core stability exercises, and functional mobility training. Sessions occur 3-4 times per week, 45-60 minutes each, during hospitalization and continued as outpatient follow-up.
  Interventions: Behavioral: Traditional Physiotherapy Rehabilitation

INTERVENTIONS:
Behavioral: Task-Oriented Rehabilitation — A structured program of repetitive, purposeful practice of everyday functional tasks (see Arm description). Delivered by trained physiotherapists 3-4 times/week, 45-60 min/session. Assigned Arm(s): Experimental: Task-Oriented Rehabilitation.
  Arms: Experimental: Task-Oriented Rehabilitation
Behavioral: Traditional Physiotherapy Rehabilitation — Standard physiotherapy focusing on stretching, strength activation, balance and functional mobility exercises. Delivered 3-4 times/week, 45-60 min/session. Assigned Arm(s): Active Comparator: Traditional Physiotherapy Rehabilitation.
  Arms: Active Comparator: Traditional Physiotherapy Rehabilitation

SUMMARY:
Stroke is one of the leading causes of long-term disability worldwide, and early rehabilitation is considered crucial for improving functional recovery. Traditional physiotherapy mainly focuses on mobility, strength, and general exercises, while task-oriented rehabilitation emphasizes practicing meaningful, goal-directed activities related to daily life. This randomized controlled trial aims to evaluate the efficacy of early task-oriented rehabilitation compared to traditional rehabilitation in acute stroke patients. Patients admitted with ischemic or hemorrhagic stroke within 48 hours will be randomly assigned to either a task-oriented rehabilitation program or conventional physiotherapy. Interventions will be delivered 3-4 times per week, 45-60 minutes per session, during hospitalization and continued in outpatient follow-up. The primary outcome will be functional independence assessed at 3 months. Secondary outcomes will include stroke severity, quality of life, and patient-reported outcomes. The findings are expected to provide evidence for improving rehabilitation strategies in Egypt.

DETAILED DESCRIPTION:
Stroke represents a major health problem worldwide and is associated with long-term disability, particularly motor dysfunction of the upper and lower limbs. Early initiation of rehabilitation is believed to enhance neuroplasticity, maximize recovery, and improve independence in daily living activities. While conventional physiotherapy focuses on stretching, balance training, and strengthening exercises, task-oriented rehabilitation emphasizes practicing functional, goal-directed tasks such as reaching for objects, buttoning shirts, sit-to-stand practice, walking, and stair climbing.

This study is a randomized controlled trial including 148-158 patients with acute ischemic or hemorrhagic stroke admitted to Assiut University Hospitals within 48 hours of onset. Participants will be randomly assigned to either the experimental group (early task-oriented rehabilitation) or the control group (traditional rehabilitation). Sessions will be delivered 3-4 times per week, each lasting 45-60 minutes, both during hospital stay and follow-up in outpatient clinics.

The primary outcome is functional recovery assessed by the Fugl-Meyer Assessment and Functional Independence Measure (FIM) at 3 months. Secondary outcomes include NIH Stroke Scale, Modified Rankin Scale, Stroke Impact Scale, depression scores, and quality of life measures.

This trial is expected to provide high-quality local evidence regarding the benefits of task-oriented rehabilitation in the acute phase of stroke recovery, which may inform clinical practice and guide rehabilitation protocols in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic or hemorrhagic stroke diagnosed clinically and confirmed by imaging.
* Admission to hospital or referral to outpatient clinic within 48 hours after stroke onset.
* Age ≥ 18 years.
* Both sexes.
* Medically stable and fit for rehabilitation.

Exclusion Criteria:

* Severe stroke not suitable for rehabilitation.
* Severe comorbidities (e.g., vital organ failure, malignancy).
* Severe aphasia, or severe visual or auditory impairment interfering with training.
* Severe upper limb spasticity (Modified Ashworth Scale > 3).
* Cognitive dysfunction (MMSE < 24 for educated; < 17 for illiterate patients).
* Stroke mimics (e.g., seizures, brain tumor, CNS infection, demyelinating diseases, hypoglycemia).
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA, Motor Domain) | Baseline (pre-intervention) At hospital discharge (Day 7-14 after admission) 3 months after hospital discharge
  Stroke-specific, performance-based scale assessing motor recovery after stroke. Score range: 0-100 (higher scores = better motor function).
  Unit of Measure: Score on a scale..

SECONDARY OUTCOMES:
Stroke Impact Scale (SIS) | Baseline (pre-intervention) At hospital discharge (Day 7-14 after admission) 3 months after hospital discharge
  Patient-reported scale assessing physical, emotion, memory, communication, and social function. Score range: 0-100 (higher scores = better quality of life). Unit of Measure: score on a scale.
Modified Rankin Scale (mRS) | Baseline (pre-intervention) At hospital discharge (Day 7-14 after admission) 3 months after hospital discharge
  Global disability scale assessing degree of dependence in daily activities. Score range: 0-6 (0 = no symptoms; 6 = death).
  Unit of Measure: Score on a scale.

REFERENCES:
- [Background] Winstein CJ, Wolf SL, Dromerick AW, Lane CJ, Nelsen MA, Lewthwaite R, Cen SY, Azen SP; Interdisciplinary Comprehensive Arm Rehabilitation Evaluation (ICARE) Investigative Team. Effect of a Task-Oriented Rehabilitation Program on Upper Extremity Recovery Following Motor Stroke: The ICARE Randomized Clinical Trial. JAMA. 2016 Feb 9;315(6):571-81. doi: 10.1001/jama.2016.0276. PMID 26864411
- [Background] French B, Thomas LH, Leathley MJ, Sutton CJ, McAdam J, Forster A, Langhorne P, Price CI, Walker A, Watkins CL. Repetitive task training for improving functional ability after stroke. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD006073. doi: 10.1002/14651858.CD006073.pub2. PMID 17943883
- [Background] Winstein CJ, Stein J, Arena R, Bates B, Cherney LR, Cramer SC, Deruyter F, Eng JJ, Fisher B, Harvey RL, Lang CE, MacKay-Lyons M, Ottenbacher KJ, Pugh S, Reeves MJ, Richards LG, Stiers W, Zorowitz RD; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Jun;47(6):e98-e169. doi: 10.1161/STR.0000000000000098. Epub 2016 May 4. PMID 27145936
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Page SJ, Gater DR, Bach-Y-Rita P. Reconsidering the motor recovery plateau in stroke rehabilitation. Arch Phys Med Rehabil. 2004 Aug;85(8):1377-81. doi: 10.1016/j.apmr.2003.12.031. PMID 15295770